CLINICAL TRIAL: NCT06844773
Title: A Single-center, Prospective, Observational Cohort Study of Chemoradiotherapy in Elderly Patients with Locally Advanced Pancreatic Cancer (70+).
Brief Title: Chemoradiotherapy in Elderly Patients with Locally Advanced Pancreatic Cancer (70+).
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZSPAC-08
Record Dates: First submitted 2025-02-06; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Unresectable Locally Advanced Pancreatic Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observation group

SUMMARY:
The goal of this observational study is to learn about the therapeutic effects of chemoradiotherapy for older adults (age 70-85) with locally advanced pancreatic cancer. The main question it aims to answer is:

Does chemoradiotherapy represent an effective and safe treatment for older participants without radical surgery? Participants will sequentially receive combined chemotherapy followed by concurrent chemoradiotherapy and subsequent maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate and sign the informed consent form
* Age 70-85 years old, life expectancy > 1 year and gender is not limited
* Eastern Cooperative Oncology Group Physical Status Score (ECOG) physical state score<=1 point
* Pathological or cytological confirmation of pancreatic ductal adenocarcinoma (including IPMN malignant transformation, acinar carcinoma, etc., excluding adenosquamous cell carcinoma and neuroendocrine carcinoma)
* The clinical stage is stage III (locally advanced pancreatic cancer), and no radical surgery has been performed (bypass surgery is acceptable), or the patient has resectable pancreatic cancer, but cannot accept surgery or refuse surgery due to physical strength or concomitant diseases
* Have not received any form of anti-tumor therapy before treatment, including systemic chemotherapy, interventional chemotherapy, high-energy focused ultrasound, radiotherapy, immunotherapy, molecular targeted therapy, and anti-tumor traditional Chinese medicine therapy
* No serious hematological, cardiological, pulmonary function abnormalities and autoimmune deficiencies (refer to their respective diagnostic criteria)
* Blood routine index: white blood cell (WBC) >=3.0 × 109/L; Absolute neutrophil count (ANC) >=1.5 × 109/L; Platelets (PLT) >=100 × 109/L; hemoglobin (Hgb) >=90 g/L
* Blood biochemical indexes: AST (SGOT), ALT (SGPT) <=2.5 × upper limit of normal value (ULN); Total bilirubin (TBIL) < = ULN; Serum creatinine (CRE) <=1.5 × ULN
* Coagulation function: prothrombin time (PT), international normalized ratio (INR) <=1.5 × ULN
* Able to comply with the requirements of the study visit plan and other programs.

Exclusion Criteria:

* Accompanied by malignant tumors of other systems
* Received any form of anti-tumor therapy before treatment, including systemic chemotherapy, interventional chemotherapy, high-energy focused ultrasound, radiotherapy, immunotherapy, molecular targeted therapy, and anti-tumor traditional Chinese medicine therapy
* Have used any other non-anti-tumor research drugs within 4 weeks before treatment
* Combined with uncontrollable hypertension, diabetes, infection, etc.
* Poor compliance, unable or unwilling to sign informed consent
* Patients who are expected to be out of the observation period for 14 days or more during the treatment period.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients with locally advanced pancreatic cancer who are evaluated by imaging at Shanghai Zhongshan hospital, aged between 70 and 85 years old, will be screened and enrolled after discussion by the ZSPAC multidisciplinary expert committee.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
1-year survival rate | From the date of first therapy administration to one year later
  To observe whether the 1-year survival rate of elderly patients with locally advanced pancreatic cancer treated with sandwich-like chemoradiotherapy modality was comparable to that of the historical data of the general adult population.

SECONDARY OUTCOMES:
Toxicity and side effects and tolerability assessment | From the date of first therapy administration to within 90 days, up to 24 months
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTCAE Version 5.0.
event-free survival throughout the enrolled subject population | From the date of first therapy administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  Survival time from the start of therapy administration to the date of first documented progression or the date of death
the proportion of participants that completed chemoradiotherapy | From the date of first enrollment to the date of completion of follow-up of the last patient, up to 24 months.
the proportion ofparticipants that completed all planned courses | From the date of first enrollment to the date of completion of follow-up of the last patient, up to 24 months.
Objective response rate (ORR) tumor target lesions in the entire subject population all planned courses | From the date of first therapy administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  ORR is defined as the percentage of patients who achieve complete response (CR) or partial response (PR) based on the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
Disease control rate (DCR) of tumor target lesions in the entire subject population all planned courses | From date of first therapy administration until the date of first documented progression or date of death from any cause, whichever occurs first, assessed up to 24 months.
  DCR is defined as the percentage of patients who achieved CR, PR and stable disease (SD), and will be evaluated based on RECIST 1.1 and the irRECIST criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No